CLINICAL TRIAL: NCT06477991
Title: The Efficacy of Watch and Wait Strategy or Surgery After Neoadjuvant Immunotherapy for Locally Advanced Colorectal Cancer With dMMR/MSI-H Guided by MRD Dynamic Monitoring(WINDOW): A Single-center, Open-label, Prospective, Phase II Clinical Trial.
Brief Title: The Efficacy of Watch and Wait Strategy or Surgery After Neoadjuvant Immunotherapy for Locally Advanced Colorectal Cancer With dMMR/MSI-H Guided by MRD Dynamic Monitoring: A Single-center, Open-label, Prospective, Phase II Clinical Trial.
Acronym: WINDOW
Status: Recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xuan Zhang, associate senior doctor, Yunnan Cancer Hospital
Other Study IDs: YJZ2023-15
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Clinical Complete Response Rate With Negative MRD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tireilizumab（PD-1 inhibitor） — Neoadjuvant immunotherapy phase :
  1. Pharmaceuticals: Tireilizumab: 200mg, intravenous infusion, Q3W, at least 4 cycles, the number of specific neoadjuvant immunotherapy cycles was determined according to the results of MRD dynamic monitoring.
  2. MRD dynamic monitoring time node: dynamic monitoring at the initial diagnosis and after the fourth cycle of neoadjuvant immunotherapy. Blood monitoring points were 1-2 weeks after immunotherapy. If the two consecutive MRDs were negative, the watch and wait strategy was adopted. If the MRD was still positive after 8 cycles of neoadjuvant immunotherapy, surgical treatment was performed.

SUMMARY:
This study is a single arm, single center, phase II, prospective clinical study aimed at exploring the effectiveness and safety of watch and wait strategy guided by dynamic minimal disease residual (MRD) monitoring to achieve clinical complete response after neoadjuvant immunotherapy for locally advanced colorectal cancer with deficient mismatch repair/ microsatellite instability-high (dMMR/MSI-H).

ELIGIBILITY:
Inclusion Criteria:

* ( 1 ) Disease characteristics 1. Histologic confirmation for colorectal adenocarcinoma; 2．Immunohistochemical identified as dMMR and/or pCR and/or NGS detection for MSI-H; 3．According to UICC/AJCC TNM staging system (in 2017 version 8) assessment for locally advanced colorectal cancer (II - III, namely cT3-4 and/or N + ）； 4.* clinical staging methods: colon CT staging, approved by pelvic magnetic resonance imaging (MRI) and the rectum rectum cavity ultrasound combined with staging, 5．No signs of intestinal obstruction;Or intestinal obstruction after proximal colon obstruction has been relieved after colostomy surgery; 6．No distant metastasis was confirmed by comprehensive examination (distant organs or (and) the distant lymph node metastasis); ( 2 ) Previous treatment 1．No colorectal cancer surgery before; 2. No previous chemotherapy or radiotherapy ; 3. had not received biological treatment ; 4. Previous endocrine therapy : no restriction.

Exclusion Criteria:

* 1.Immunohistochemistry of tumor biopsy specimens suggested pMMR or microsatellite instability detection suggested MSS ; 2. Chronic hepatitis B or C ( high-copy viral DNA ) with a history of HIV infection or active phase ; 3.Autoimmune diseases ; 4.Other active clinical severe infections ( > NCI-CTC3.0 version ) ; 5. patients with clinical stage I ; 6.Preoperative evidence of distant metastasis ; 7. cachexia, organ dysfunction ; 8. Have a history of pelvic or abdominal radiotherapy ; 9. Patients whose seizures require treatment ( e.g. steroids or antiepileptic treatment ) ; 10.5 years have a history of other malignant tumors, except for cured cervical carcinoma in situ or skin basal cell carcinoma ; 11. Chronic inflammatory bowel disease, intestinal obstruction ; 12. Drug abuse and medical, psychological or social conditions may interfere with patient participation in the study or have an impact on the evaluation of the results of the study ; 13.Known or suspected allergies to the study drug or any drug related to this test ; any unstable condition or condition that may endanger patient safety and compliance ;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ( 1 ) Patient characteristics
  1. Age : 18-75 years old ;
  2. Physical status score : ECOG 0-1 ;
  3. Life expectancy : more than 2 years ;
  4. hematology : WBC > 4000 / mm3 ; pLT > 100000 / mm3 ; hb should be > 10g / dL in principle ; chronic anemia ( hemoglobin < 10.0 g / dL ) is not an exclusion criterion but should be corrected by blood transfusion before surgery and chemotherapy. If hemoglobin remains low after transfusion, surgery and chemotherapy can be decided by surgical and medical teams.
  5. Liver function : SGOT and SGPT were less than 1.5 times of normal value ; bilirubin less than 1.5 mg / dL ;
  6. Renal function : creatinine < 1.8mg / dL ;
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response rate with negative MRD | 2023/10/30-2026/10/30
  Clinical complete response rate with negative MRD

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-07-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT06477991/Prot_000.pdf
  • Informed Consent Form (2023-07-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT06477991/ICF_001.pdf